CLINICAL TRIAL: NCT01252004
Title: French Observatory Syndromes Tako-Tsubo
Acronym: OFSETT
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Jean-Jacques DUJARDIN, Professor, French Cardiology Society
Other Study IDs: OFSETT
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Necrosis; Tako Tsubo Syndromes
Keywords: Left ventricular ballooning
MeSH Terms: conditions — Myocardial Infarction; Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TT Syndrome: Will be included over a period of one year, prospectively, all patients newly diagnosed

SUMMARY:
Tako Tsubo syndrome (TTS) is characterized by the occurrence in the context of mental or physical stress, a clinical and ECG of acute myocardial infarction without significant coronary artery stenosis, accompanied by a disorder Acute, reversible left ventricular who takes on a characteristic apical ballonnisation evoking the image of a Japanese octopus trap called Tako (octopus) tsubo (jar). Pathophysiology of unknown changes immediate life-threatening prognosis is often good in the longer term.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* allowed for an array of myocardial necrosis on clinical and electro cardiographic
* having a left ventricular ballooning echo cardiography, MRI or ventriculographic with normal coronary angiogram.

Exclusion Criteria:

* Absence of left ventricular ballooning and / or presence of coronary lesions on angiography
* Refusal by the patient to participate in the observatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed for a Tako-Tsubo Syndrome. Recruitment will be from the centers of coronary angiography and coronary angioplasty in high volume.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Psychological events | 1 day
  Study of psychological events that triggered the event by using the stress scale of the Canadian Association for Mental Health

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Dujardin, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CH Douai, Douai, France

REFERENCES:
- [Background] Kurisu S, Sato H, Kawagoe T, Ishihara M, Shimatani Y, Nishioka K, Kono Y, Umemura T, Nakamura S. Tako-tsubo-like left ventricular dysfunction with ST-segment elevation: a novel cardiac syndrome mimicking acute myocardial infarction. Am Heart J. 2002 Mar;143(3):448-55. doi: 10.1067/mhj.2002.120403. PMID 11868050
- [Background] Tsuchihashi K, Ueshima K, Uchida T, Oh-mura N, Kimura K, Owa M, Yoshiyama M, Miyazaki S, Haze K, Ogawa H, Honda T, Hase M, Kai R, Morii I; Angina Pectoris-Myocardial Infarction Investigations in Japan. Transient left ventricular apical ballooning without coronary artery stenosis: a novel heart syndrome mimicking acute myocardial infarction. Angina Pectoris-Myocardial Infarction Investigations in Japan. J Am Coll Cardiol. 2001 Jul;38(1):11-8. doi: 10.1016/s0735-1097(01)01316-x. PMID 11451258
- [Background] Sharkey SW, Lesser JR, Zenovich AG, Maron MS, Lindberg J, Longe TF, Maron BJ. Acute and reversible cardiomyopathy provoked by stress in women from the United States. Circulation. 2005 Feb 1;111(4):472-9. doi: 10.1161/01.CIR.0000153801.51470.EB. PMID 15687136
- [Background] Parodi G, Del Pace S, Carrabba N, Salvadori C, Memisha G, Simonetti I, Antoniucci D, Gensini GF. Incidence, clinical findings, and outcome of women with left ventricular apical ballooning syndrome. Am J Cardiol. 2007 Jan 15;99(2):182-5. doi: 10.1016/j.amjcard.2006.07.080. Epub 2006 Nov 14. PMID 17223415
- [Background] Gianni M, Dentali F, Grandi AM, Sumner G, Hiralal R, Lonn E. Apical ballooning syndrome or takotsubo cardiomyopathy: a systematic review. Eur Heart J. 2006 Jul;27(13):1523-9. doi: 10.1093/eurheartj/ehl032. Epub 2006 May 23. PMID 16720686
- [Background] El Mahmoud R, Mansencal N, Pilliere R, Leyer F, Abbou N, Michaud P, Nallet O, Digne F, Lacombe P, Cattan S, Dubourg O. Prevalence and characteristics of left ventricular outflow tract obstruction in Tako-Tsubo syndrome. Am Heart J. 2008 Sep;156(3):543-8. doi: 10.1016/j.ahj.2008.05.002. Epub 2008 Jul 7. PMID 18760139
- [Background] Eitel I, Behrendt F, Schindler K, Kivelitz D, Gutberlet M, Schuler G, Thiele H. Differential diagnosis of suspected apical ballooning syndrome using contrast-enhanced magnetic resonance imaging. Eur Heart J. 2008 Nov;29(21):2651-9. doi: 10.1093/eurheartj/ehn433. Epub 2008 Sep 27. PMID 18820322
- [Result] Yayehd K, N'da NW, Belle L, Bataille V, Hanssen M, Leddet P, Aupetit JF, Commeau P, Filippi E, Georges JL, Albert F, Range G, Meimoun P, Marcaggi X, Baleynaud S, Nallet O, Dibie A, Barnay C, Jouve B, Legrand M, Cattan S, Mulak G, Simon T, Danchin N, Dujardin JJ; OFSETT investigators. Management of Takotsubo cardiomyopathy in non-academic hospitals in France: The Observational French SyndromEs of TakoTsubo (OFSETT) study. Arch Cardiovasc Dis. 2016 Jan;109(1):4-12. doi: 10.1016/j.acvd.2015.08.004. Epub 2015 Oct 23. PMID 26507532